CLINICAL TRIAL: NCT04530045
Title: Target Attainment of TDM-guided Continuous Infusion of Piperacillin/Tazobactam and Cefepim in Critically Ill Patients: a Prospective Observational Study
Brief Title: Target Attainment of TDM-guided Infusion of Piperacillin/Tazobactam and Cefepim in Critically Ill Patients
Acronym: DOSATB
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/DOSATB-NOVY/YB
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness; Antibiotic Toxicity; Sepsis; Septic Shock
Keywords: therapeutic drug monitoring
MeSH Terms: conditions — Critical Illness; Sepsis; Shock, Septic | interventions — Cefepime

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill patients: Critically ill patients receiving continuous infusion of piperacillin/tazbactam or cefepim and dosage of plasma concentration of the B lactam administered
  Interventions: Other: dosage of concentration of piperacillin and cefepim

INTERVENTIONS:
Other: dosage of concentration of piperacillin and cefepim — Dosage of total plasma concentration of piperacillin and cefepim at different timepoints

SUMMARY:
Although alternative dosing strategies can improve antimicrobial exposure in critically ill patients, the high PK variability in this population means that some may still receive sub-optimal antibiotic exposure leading to unfavourable clinical outcomes.

Therapeutic drug management (TDM) guided dosing is the only safe and effective way to ensure that all critically ill patients achieve therapeutic antimicrobial exposures and to minimise the likelihood of toxicity.

For experts, TDM should be a standard of care, in particular for β-lactams. Nevertheless, because of the assay method for β-lactams and the need for bioanalytical experts, delays in obtaining results frequently occurred. These barriers, combined with difficulties in the interpretation of TDM results, need to be addressed in order to increase its routine utilization. Consequently, study aiming at identify which subgroup of patients or infection are more likely to benefit from TDM are urgently warranted This prospective observational study aimed at evaluating target attainment of piperacillin/tazobactam (PIP/TAZ) and cefepim (CEF) with the use of a Therapeutic Drug Monitoring (TDM) in critically patients during the routine care

ELIGIBILITY:
Inclusion Criteria:

* Minimun age limits 18 years
* Critically ill patient receiving piperacillin or cefepim administered continuously

Exclusion Criteria:

* Beta lactam allergy
* Pregnancy
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the surgical intensive care unit whatever the reason of admission and who received piperacilin or cefepim with a TDM for sepsis or septic shock during their stay.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
to determine the percentage of patients who met the PK/PD targets at 24 hours | Day 1
  PK/PD target was defined as follows:
  Concentration of piperacillin or cefepim between a lower and a upper limit:
  * The lower limit was defined as estimated free concentration above 4 times the epidemiological cut-off value of suspected bacteria
  * The upper limit was based on known limit of neurotoxicity, namely 35 and 160 mg/L for cefepim and piperacillin, respectively
  Consequently :
  * for piperacillin : the PK/PD target is considered to be reach if the free concentration of PIPERACILLIN/TAZOBACTAM is between 32 and 160 mg/l
  * for cefepim : the PK/PD target is considered to be reach if the free concentration of CEFEPIM is between 4 and 35 mg/l

SECONDARY OUTCOMES:
to determine the percentage of patients who met the PK/PD targets "exposure" at 24 hours | Day 1
  PK/PD target "exposure" take into account only the the lower limit was defined as estimated free concentration above 4 times the epidemiological cut-off value of suspected bacteria
  Consequently :
  * for piperacillin : the PK/PD target is considered to be reach if the free concentration of PIPERACILLIN/TAZOBACTAM is above 32 mg/l
  * for cefepim : the PK/PD target is considered to be reach if the free concentration of CEFEPIM is above 4 mg/l
factors associated with target attainment at day 1 | Statistical analysis after 2 years of inclusion
  effect of age on antibiotic concentration
factors associated with target attainment at day 1 | Statistical analysis after 2 years of inclusion
  effect of renal clearance on antibiotic concentration
factors associated with target attainment at day 1 | Statistical analysis after 2 years of inclusion
  effect of presence of septic shock on antibiotic concentration
factors associated with dose changing | Statistical analysis after 2 years of inclusion
  effect of presence of septic shock on number of dose changing after analyse of antibiotic concentration
factors associated with dose changing | Statistical analysis after 2 years of inclusion
  effect of renal clearance on number of dose changing after analyse of antibiotic concentration

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel NOVY, Principal Investigator — Central Hospital, Nancy, France
Locations (2):
- France (2):
  - Emmanuel NOVY, Vandœuvre-lès-Nancy, Lorraine
  - Central Hospital, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No